CLINICAL TRIAL: NCT01341028
Title: Effects of the Resection of the Gastric Fundus on the Secretion of Ghrelin, Peptide-YY, Glucagon-like Peptide-1 and Insulin Secretion in Morbidly Obese Patients Undergoing Laparoscopic Roux-en-Y Gastric Bypass
Brief Title: Gut Hormones After Roux-en-Y Gastric Bypass (RYGBP) Plus Gastric Fundus Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Theodore K. Alexandrides, Professor of Medicine, University of Patras School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RYGBPFR001
Record Dates: First submitted 2011-04-18; First posted 2011-04-25 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2007-02

CONDITIONS: Morbid Obesity
Keywords: weight loss; appetite; ghrelin; PYY; GLP-1; insulin; laparoscopic; Roux-en-Y gastric bypass; gastric fundus resection
MeSH Terms: conditions — Obesity, Morbid; Weight Loss; Insulin Resistance | interventions — Gastric Bypass

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Roux-en-Y gastric bypass (LRYGBP) (Active Comparator): Twelve subjects underwent laparoscopic Roux-en-Y gastric bypass
  Interventions: Procedure: Roux-en-Y gastric bypass (LRYGBP)
- LRYGBP plus gastric fundus resection (Experimental): Twelve patients underwent laparoscopic Roux-en-Y gastric bypass plus gastric fundus resection
  Interventions: Procedure: LRYGBP+gastric fundus resection

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass (LRYGBP) — Twelve patients underwent laparoscopic Roux-en-Y gastric bypass
  Other Names: LRYGBP
  Arms: Roux-en-Y gastric bypass (LRYGBP)
Procedure: LRYGBP+gastric fundus resection — Twelve patients underwent laparoscopic Roux-en-Y gastric bypass and gastric fundus resection
  Arms: LRYGBP plus gastric fundus resection

SUMMARY:
* Laparoscopic Roux-en-Y gastric bypass (LRYGBP) is considered a combination of restriction-malabsorption procedure and one of the most common operative procedures implemented.
* Over the last years increasing evidence suggests that the beneficial effects of bariatric operations might be related to the suppression of appetite caused by the release of the anorectic gut hormones such as peptide-YY (PYY) and glucagon-like peptide-1 (GLP-1)by the L cells of the distal gut and the suppression of the orexigenic hormone ghrelin released by the stomach.Obese people have a blunted rise in PYY and GLP-1 after a meal, possibly resulting in impaired satiety and hence greater food intake.
* In the present study the investigators sought to evaluate the effects of the resection of the gastric fundus, the main source of ghrelin production, on the secretion of ghrelin, PYY, GLP-1 and insulin and in addition on glucose levels, appetite and weight loss, in morbidly obese patients undergoing laparoscopic Roux-en-Y gastric bypass.

DETAILED DESCRIPTION:
Twenty four patients were included prospectively in the study. After randomization, 12 patients underwent LRYGBP and 12 LRYGBP plus gastric fundus resection (LRYGBP+FR).

All human studies were performed according to the principles of the Declaration of Helsinki. The local Research and Ethics Commitee at the University Hospital of Patras approved the study. Written informed consent was obtained from all patients.

All the operations were performed by the same surgeon laparoscopically. The RYGBP procedures were performed creating a small isolated lesser curve-based gastric pouch (20 ± 5 ml) and a 150cm Roux limb. The gastroenteroanastomosis was conducted with a 25 mm circular stapler. The dissection of the fundus of the stomach in the (LRYGBP+FR) group was done with the use of EndoGia No 60.

The subjects were studied before and at 3, 6 and 12 months after the operation. All the patients underwent an oral glucose tolerance test (OGTT) with 75 g glucose, preoperatively. In addition, venous blood was collected after an overnight 12 hour fast and 30, 60 and 120 min after the administration of a 300 kcal mixed meal.The meal was consumed in ten minutes and consisted of 18% protein, 55% carbohydrate and 27% fat (Resource energy drink, Nestle Nutrition, France). Plasma levels of PYY, GLP-1, ghrelin and insulin were determined at every time point of the study. All patients underwent complete clinical evaluation during follow-up including nutritional, behavioral and anthropometric parameters. Visual analogue scales (VAS) were used to measure hunger, nausea, fullness and aversion to food, before and 30, 60 and 120 min after the consumption of the meal. Weight loss evaluation was based on postope¬rative body weight, body mass index (BMI) and % excess weight loss (EWL %).

Insulin resistance was approximated using the homeostatic model assessment for insulin resistance (HOMA IR). The following formula was used in its calculation:

HOMA IR = (fasting glucose [mmole] /lt X fasting insulin [μU/ml])/22.5). The insulinogenic index, a commonly used indicator of pancreatic β-cell function, was calculated as the ratio of increment of insulin concentrations to that of glucose concentrations at 30 minutes after meal ingestion (Δ [ins30 - ins0] / Δ [Glu30 -Glu0]).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index higher than 40 kg/m2

Exclusion Criteria:

* pregnancy
* diabetes mellitus
* substance abuse
* chronic medical or psychiatric illness
* previous gastrointestinal surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The effects of the resection of the gastric fundus on the secretion of ghrelin, PYY, GLP-1 and insulin. | The outcome was assessed 12 months after the operation
  The effect on the secretion of ghrelin, PYY, GLP-1 and insulin

SECONDARY OUTCOMES:
The effects of the resection of the gastric fundus on glucose levels, appetite and weight loss | At 12 months after the operation
  The effect of fundus resection on glucose levels, appetite and weight loss was assessed 12 months after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Theodore K Alexandrides, Principal Investigator — Professor of Medicine, School of Medicine, University of Patras
Locations (1):
- University Hospital of Patras, Rio, Achaia, Greece